CLINICAL TRIAL: NCT04026529
Title: Improving Exercise Capacity in Chronic Obstructive Pulmonary Disease Patients Through Uphill Walking
Brief Title: Uphill Walking as Exercise for COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: E3294-P; 1I21RX003294-01 (NIH)
Record Dates: First submitted 2019-07-18; First posted 2019-07-19 (Actual); Results first posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: pulmonary rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Cross-sectional design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- walking at incline (Experimental): Subjects will walk on treadmill at slope and speed to equal 60% of their peak work rate as determined on baseline cardiopulmonary exercise test.
  Interventions: Other: walking on incline or walking at increasing speed

INTERVENTIONS:
Other: walking on incline or walking at increasing speed — Subjects will be prepared for data collection by wearing a form-fitting suit (i.e., wrestling singlet) and obtaining height and body weight. Retro-reflective markers will be placed bilaterally on anatomical locations of the feet, legs, and hips.
  Subjects will be outfitted with the portable metabolic cart and oximeter as in the previous visit. One of two treadmill trials will be performed: 1) at the speed and 2) at the slope +speed determined in the previous visit. Trial order will be randomized among subjects and across visits 3 & 4. For each trial, subjects will be asked to walk on a treadmill for up to 6 minutes. Speed or slope will be increased every 30 seconds and they will be asked to walk for one minute at that speed or slope.

SUMMARY:
This study is designed to provide preliminary information regarding how to improve pulmonary rehabilitation for persons with chronic obstructive pulmonary disease (COPD). Pulmonary rehabilitation is an exercise program for COPD patients that is recommended and benefits some, but not all, patients. The question being studied in this trial is whether walking on an incline might be better than walking on faster on a flat surface in training muscles so that patients might be less short of breath with exercise.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a major cause of morbidity and mortality and presents an important healthcare problem, especially for Veterans. Prevalence of COPD in the Veteran population ranges from 33%-43%, a higher prevalence than among the general population of the United States. COPD patients experience diminished exercise capacity. A significant portion of this limitation in exercise capacity is due to dynamic hyperinflation and dyspnea. Humans demonstrate a coupled relationship between walking and breathing. The investigators' preliminary data indicates that patients with COPD demonstrate an abnormal coupling pattern compared to those without COPD, using one stride for one breath, even at speeds outside of their self-selected walking pace. Current pulmonary rehabilitation relies on increasing intensity of exercise through accelerated walking. Based on coupling patterns in patients with COPD, increasing speed leads to an increase in respiratory rate, dynamic hyperinflation, and dyspnea, thus limiting exercise time. The goal of this proposed project is to investigate, in Veteran COPD patients, the effect of walking faster vs. walking on a slope on dynamic hyperinflation and dyspnea, oxygen uptake and dead space, and walking and breathing coupling. The investigators hypothesize that walking on a slope will alter breathing and walking coupling, lower respiratory rates, and reduce dynamic hyperinflation and associated dyspnea. The investigators predict that walking on a slope will permit an increase in oxygen uptake and a decrease in dead space in patients with COPD as compared to accelerated walking speeds. These hypotheses will be tested through three aims: 1) Identify differences in dynamic hyperinflation and dyspnea; 2) Compare differences in respiratory rate, oxygen uptake, and lung dead space; 3) Determine the complexity of walking and breathing coupling ratios. In this cross-sectional study, Veterans with COPD will be recruited and screened using a cardiopulmonary exercise test. A total of 25 eligible Veterans will be enrolled through stratified sampling of disease severity. The time course of work rate will be calculated from the cardiopulmonary exercise test. The speed and slope that corresponds to 60% of peak work rate will be used. An additional constant work rate test will be given using increases in speed with a level treadmill to determine the speed that elicits oxygen uptake comparable to the sloped walking test. Subjects will be asked to perform two experimental trials (walking faster vs. walking on a slope) at 60% peak work rate. Measures of dynamic hyperinflation, dyspnea, oxygen uptake, dead space, and coupling will be recorded during all walking trials. Possible covariates will also be collected. The investigators anticipate that dynamic hyperinflation and dyspnea will be reduced in patients with COPD due to slower walking and slower respiratory rates during sloped walking as compared to faster level walking. It is expected that this will be influenced by the complexity in breathing and walking coupling ratios. The investigators' multidisciplinary team will provide combined expertise from several disciplines and is uniquely qualified to complete the aims proposed. Results from this feasibility and acceptability study will set the stage for a rigorous, well-powered, full Merit award outcome study evaluating the effectiveness of a slope-based training regimen as part of rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Veterans from all sex/gender, race, and ethnicity will be recruited
* All subjects will undergo post-bronchodilator spirometry and be clinically stable
* All subjects must have documented FEV1/FVC ratio of <0.7, and between 30% to 80% FEV1% predicted
* If subjects have non-qualifying spirometry, they will not be screened further
* Subjects with qualifying spirometry will be screened further
* Potential subjects must have a BMI of less than 35 kg/m2 and must be free from co-morbidities that may affect walking patterns

  * e.g., peripheral arterial disease, diabetes, low back pain

Exclusion Criteria:

* Confounding effects such as neurological, musculoskeletal, or metabolic disease
* Subjects taking medications that alter mood or metabolic demand will be excluded
* All potential subjects must be cleared for participation by a physician after undergoing a cardiopulmonary exercise test
* Require an O2 mask during rest or activity

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debra J. Romberger, MD, Principal Investigator — Omaha VA Nebraska-Western Iowa Health Care System, Omaha, NE
Locations (1):
- Omaha VA Nebraska-Western Iowa Health Care System, Omaha, NE, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Walking at Incline or Speed: Subjects will walk on treadmill at slope and speed to equal 60% of their peak work rate as determined on baseline cardiopulmonary exercise test.
  Walking on incline or walking at increasing speed: Subjects will be prepared for data collection by wearing a form-fitting suit (i.e., wrestling singlet) and obtaining height and body weight. Retro-reflective markers will be placed bilaterally on anatomical locations of the feet, legs, and hips.
  Subjects will be outfitted with the portable metabolic cart and oximeter as in the previous visit. One of two treadmill trials will be performed: 1) at the speed and 2) at the slope +speed determined in the previous visit. Trial order will be randomized among subjects and across visits 3 & 4. For each trial, subjects will be asked to walk on a treadmill for up to 6 minutes. Speed or slope will be increased every 30 seconds and they will be asked to walk for one minute at that speed or slope.
Period: Overall Study
Arm/Group | Walking at Incline or Speed
Started | 8 (10/21/2020)
Completed | 8 (09/30/2022)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Walking at Incline or Speed
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.25 (3.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8
Participants have COPD. [Count of Participants; unit: Participants] — COPD defined by spirometry with FEV1/FVC ratio less than 70%
  Participants | 8

OUTCOME MEASURES:

1. Primary Outcome: Dyspnea
Description: Perceived dyspnea: Breathlessness will be measured based on a 0 to 10-point Borg scale at the end of the treadmill trials. 0 on scale is no breathlessness and 10 is maximal breathlessness
Time Frame: Visits were assessed at pre-specified randomized slope/speed treadmill intervals, with each visit scheduled to occur within one week of the previous visit, all taking place within a 6-week period following enrollment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Walking at Incline or Speed
Number analyzed (Participants) | 8
score on a scale
  slope visit, randomized either 3 or 4 | 9.62 (2.55)
  speed visit, randomized either 3 or 4 | 9.12 (3.04)

2. Other Pre Specified Outcome: Dynamic Hyperinflation
Description: Dynamic hyperinflation will be assessed by inspiratory capacity through pre- and post-walking trial resting spirometry. Dynamic hyperinflation will be considered to be present when inspiratory capacity values decrease after walking trials when compared to resting values.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of tidal volume/lung capacity
Arm/Group | Walking at Incline or Speed
Number analyzed (Participants) | 8
Percentage of tidal volume/lung capacity
  slope visit randomized either 3rd or 4th visit | 0.21 (0.61)
  speed visit randomized either 3rd or 4th visit | -0.11 (0.42)

3. Other Pre Specified Outcome: Respiratory Rate
Description: Respiratory rate will be analyzed using motion capture markers on the chest. With custom computer code, the markers will be identified to model a sphere. The volume of the sphere will be recorded over time. As the volume increases and decreases, respiratory flow will be identified, and respiratory rate can be calculated.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: breath per minute
Arm/Group | Walking at Incline or Speed
Number analyzed (Participants) | 8
breath per minute
  slope visit, randomized either 3rd or 4th visit | 27.49 (6.79)
  speed visit, slope visit, randomized either 3rd or 4th visit | 26.5 (6.34)

4. Other Pre Specified Outcome: Percentage of Time in Which the Most Common Ratio of Coupling Was Detected
Description: The laboratory is equipped with a 17-camera, digital motion capture system (Motion Analysis Corp., Santa Rosa, CA; 120Hz) to allow for collection of three-dimensional marker positions in real time.
  The breathing cycle will be determined based on the movement of markers placed on the chest, while the gait cycles will be identified using locomotor data derived from heel markers, focusing on heel contact events.
  Coupling is often quantified as frequency coupling. Frequency coupling refers to how many heel strikes occur within a single cycle of respiration (one inhalation to the next).
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Walking at Incline or Speed
Number analyzed (Participants) | 8
percentage of time
  slope visit randomized either 3rd or 4th visit | 51.08 (24.67)
  speed visit randomized either 3rd or 4th visit | 74.13 (14.43)

5. Other Pre Specified Outcome: Oxygen Uptake
Description: Heart rate and pulmonary gas exchange analysis will be recorded on a breath-by-breath basis. This will provide an accurate measure of pulmonary gas exchange, including oxygen uptake, i.e. VO2, . Steady-state VO2 while walking will be averaged and normalized to standing metabolic rate.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Walking at Incline or Speed
Number analyzed (Participants) | 8
ml/kg/min
  slope visit randomized either 3rd or 4th visit | 14.16 (3.50)
  speed visit randomized either 3rd or 4th visit | 15.28 (4.45)

6. Other Pre Specified Outcome: Lung Dead Space
Description: Dead space: Tidal volume and expired carbon dioxide will be measured using the same equipment as oxygen uptake above. Partial pressure of arterial carbon dioxide will be measured using a transcutaneous sensor.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Walking at Incline or Speed
Number analyzed (Participants) | 8
ml
  slope visit randomized either 3rd or 4th visit | 0.48 (0.19)
  speed visit randomized either 3rd or 4th visit | 0.51 (0.18)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Walking at Incline or Speed
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

LIMITATIONS AND CAVEATS:
Study enrollment impacted by COVID-19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-14): https://cdn.clinicaltrials.gov/large-docs/29/NCT04026529/Prot_SAP_001.pdf
  • Informed Consent Form (2021-11-02): https://cdn.clinicaltrials.gov/large-docs/29/NCT04026529/ICF_000.pdf